CLINICAL TRIAL: NCT00514189
Title: Feasibility Study of Acute Myelogenous Leukemia mRNA Plus Lysate Loaded Dendritic Cell Vaccines
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated early due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0379
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: Acute Myelogenous Leukemia; Leukemia; Autologous Dendritic Cells; Vaccine; AML; mRNA
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Dendritic Cells (Experimental)
  Interventions: Biological: Autologous Dendritic Cells

INTERVENTIONS:
Biological: Autologous Dendritic Cells — The first vaccination will be given once your blood counts have recovered from the final dose of chemotherapy. The remaining 3 vaccinations will be given every 28 days (+/- 7 days).
  Other Names: DCs

SUMMARY:
Primary Objectives:

1. To determine the feasibility of delivering autologous dendritic cells (DCs) loaded with acute myelogenous leukemia (AML) lysate plus messenger RNA (mRNA) to AML patients following consolidation therapy.
2. To determine the toxicity of autologous DCs loaded with AML lysate plus mRNA.
3. To quantitate immune responses in patients who receive autologous DCs loaded with AML lysate plus mRNA.

Secondary Objectives:

1. To evaluate minimal residual disease following DC therapy using the polymerase chain reaction assay for the Wilm's Tumor-1 gene.
2. To asses the disease-free and overall survival of AML patients who receive the autologous DCs loaded with AML lysate plus mRNA.

DETAILED DESCRIPTION:
Patient Consent: Arm 1 - Standard-Dose Consolidation

The vaccine will be made from your AML cells which will be killed, frozen, and stored away when you start the study. When you go into remission, researchers will take your normal blood cells and culture them in the laboratory until they become "dendritic cells." Researchers will then thaw your tumor cells and load parts of them into the dendritic cells and inject the mixture. This type of vaccine will hopefully encourage your immune system to prevent later relapse of your disease.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Blood (about 1 tablespoon) will be drawn to make sure you do not have an infection with HIV/AIDS. If you do, you will not be eligible for this study.

If you are found to be eligible to take part in this study, AML cells will be collected from your blood through a vein in your arm. A blood separator device called an apheresis machine will be used. Each apheresis procedure takes about 3-5 hours. It is similar to donating platelets to a blood bank. During the procedure the blood with tumor cells will be removed and then returned through a second line in the other arm. You may have bone marrow aspirations instead with general anesthesia, usually lasting up to 3 hours. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle. The AML cells collected by either the apheresis or bone marrow collection procedure will be used later to make the vaccine in the M. D. Anderson Cell Therapy Laboratory where they will be frozen and stored until it is time to make the vaccine.

After the AML cells are collected, you will start receiving your induction and consolidation chemotherapy treatment. This treatment is standard of care and is not directly related to your participation in this study. After your first cycle of consolidation treatment, a bone marrow biopsy will be done to find out if you are in complete remission. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. If you are in complete remission then you will have your normal blood stem cells collected, which will be used to make the vaccine. All of the normal stem cells will be collected with the same apheresis machine used to collect tumor cells. Beginning 5 days before the first collection, you will receive daily injections under the skin of granulocyte colony stimulating factor (G-CSF). These are given to increase the number of normal stem cells available for collection. On Days 5 and 6 of G-CSF treatment, your normal stem cells will be collected. They will be taken to the M. D. Anderson Cell Therapy Laboratory where they will be frozen and stored until it is time to make the vaccine.

After you complete the apheresis procedure to collect normal cells, you will continue consolidation therapy (typically 3-5 cycles). The vaccine will be made with your previously frozen cells. Once thawed, a machine called the CliniMACS will be used to isolate the cells from your blood that will be grown into the vaccine during an 8-day procedure.

After the last consolidation cycle, you will begin to receive 4 monthly injections of the vaccine. The first vaccination will be given once your blood counts have recovered from the final dose of chemotherapy. The remaining 3 vaccinations will be given every 28 days (+/- 7 days). Once it is ready, each vaccine will be injected into a lymph node in your groin. A special machine called a sonogram (typically used to look at babies in the womb) will be used to painlessly locate exactly where the injection should go.

About 3-7 days after each vaccine, about 4 tablespoons of your blood will be drawn to measure the immune reaction to the vaccine. At that time you will also have a skin test performed to look for the presence or absence of an immune reaction to the vaccine. This will be done with a small injection under the skin on your forearm. About 48 hours later, researchers will measure the area around the injection for redness, which would be a sign that your immune system is reacting to the vaccine.

After you have received all 4 vaccines, you will be seen in the clinic yearly to evaluate how you tolerated the vaccines.

Routine long-term follow-up exams will be performed by your leukemia doctor as per standard of care.

This is an investigational study. The vaccines are not commercially available and only authorized for use in research. A total of 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

Patient Consent: Arm 2 - Autologous Peripheral Blood Progenitor Cell Consolidation

The vaccine will be made from your AML cells which will be killed, frozen, and stored away when you start the study. When you go into remission, researchers will take your normal blood cells and culture them in the laboratory until they become "dendritic cells." Researchers will then thaw your tumor cells and load parts of them into the dendritic cells and inject the mixture. This type of vaccine will hopefully encourage your immune system to prevent later relapse of your disease.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Blood (about 1 tablespoon) will be drawn to make sure you do not have an infection with HIV/AIDS. If you do, you will not be eligible for this study.

If you are found to be eligible to take part in this study, AML cells will be collected from your blood through a vein in your arm. A blood separator device called an apheresis machine will be used. Each apheresis procedure takes about 3-5 hours. It is similar to donating platelets to a blood bank. You may have bone marrow aspirations instead with general anesthesia, usually lasting up to 3 hours. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle. The AML cells collected by either the apheresis or bone marrow collection procedure will be used later to make the vaccine in the M. D. Anderson Cell Therapy Laboratory where they will be frozen and stored until it is time to make the vaccine.

After the AML cells are collected, you will start receiving your induction and consolidation chemotherapy treatment. This treatment is standard of care and is not directly related to your participation in this study. After your first cycle of consolidation treatment, a bone marrow biopsy will be done to find out if you are in complete remission. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. If you are in complete remission then you will have your normal blood stem cells collected, which will be used to make the vaccine. All of the normal stem cells will be collected with the same apheresis machine used to collect tumor cells. Beginning 5 days before the first collection, you will receive daily injections under the skin of granulocyte colony stimulating factor (G-CSF). These are given to increase the number of normal stem cells available for collection. On Days 5 and 6 of G-CSF treatment, your normal stem cells will be collected. They will be taken to the M. D. Anderson Cell Therapy Laboratory where they will be frozen and stored until it is time to make the vaccine.

After you complete the apheresis procedure to collect normal cells, you will continue consolidation therapy with high-dose standard busulfan and cyclophosphamide chemotherapy. You will also have an autologous peripheral blood progenitor cell transplant. The chemotherapy and transplant are standard of care.

After the chemotherapy and transplant when your blood counts have recovered, you will begin to receive 4 monthly injections of the vaccine. The vaccine will be made with your previously frozen cells. Once thawed, a machine called the CliniMACS will be used to isolate the cells from your blood that will be grown into the vaccine during an eight day procedure.

The first vaccination will be given once your blood counts have recovered from the final dose of chemotherapy. The remaining 3 vaccinations will be given every 28 days (+/- 7 days). Once it is ready, each vaccine will be injected into a lymph node in your groin. A special machine called a sonogram (typically used to look at babies in the womb) will be used to painlessly locate exactly where the injection should go.

About 3-7 days after each vaccine, about 4 tablespoons of your blood will be drawn to measure the immune reaction to the vaccine. At that time you will also have a skin test performed to look for the presence or absence of an immune reaction to the vaccine. This will be done with a small injection under the skin on your forearm. About 48 hours later, researchers will measure the area around the injection for redness, which would be a sign that your immune system is reacting to the vaccine.

After you have received all 4 vaccines, you will be seen in the clinic to evaluate how you tolerated the vaccines.

Routine long-term follow-up exams will be performed by your leukemia doctor yearly as per standard of care.

This is an investigational study. The vaccines are not commercially available and only authorized for use in research. A total of 20 patients take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated AML except patients with inv (16), t(8;21), or t (15;17) cytogenetics or AML in first relapse.
2. Patients must have >/= 2,000 circulating blasts/ul peripheral blood or >/= 50% blasts in bone marrow biopsy
3. Performance Status 0-2

Exclusion Criteria:

1. Medical, social or psychological factors which would prevent the patient from receiving or cooperating with the full course of therapy or understanding the informed consent procedure.
2. Concurrent or expected need for therapy with corticosteroids during the vaccination phase of the study.
3. History of systemic autoimmune disease
4. Positive antibody to human immunodeficiency virus
5. Patients with Acute promyelocytic Leukemia are not eligible for this study.
6. Good-risk cytogenetics which are: (inv (16), t(8;21), or t (15;17)
7. Positive Beta HCG test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to Adverse Event (AE) | Day of First Vaccination to 6 Months Follow Up After Last Patient Accrued

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org